CLINICAL TRIAL: NCT06753565
Title: Effect of L-carnitine Supplementation on Disease Activity in Rheumatoid Arthritis Patients
Brief Title: L-carnitine Supplementation in Rheumatoid Arthritis Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: German University in Cairo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RACAR
Record Dates: First submitted 2024-11-26; First posted 2024-12-31 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis; Carnitine; anti-inflammatory; anti-oxidant; ACR50%; disease activity
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Carnitine; Antirheumatic Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- l-carnitine and conventional DMARDs (Experimental): l-carnitine 500 mg ( carnitine tartrate 500 mg) two capsules twice daily for three months as add on therapy to conventional DMARDs.
  Interventions: Drug: Carnitine; Drug: Disease-modifying anti-rheumatic drugs
- placebo and conventional DMARDs (Placebo Comparator): placebo 500 mg two capsules twice daily for three months as add on therapy to conventional DMARDs.
  Interventions: Drug: Disease-modifying anti-rheumatic drugs

INTERVENTIONS:
Drug: Carnitine — It is a nutritional supplement with trade name " Carnitol®" in Egypt.
  Arms: l-carnitine and conventional DMARDs
Drug: Disease-modifying anti-rheumatic drugs — They are immunosuppressive drugs used to improve disease activity in Rheumatoid Arthritis patients . Conventional DMARDs include methotrexate (Imutrexate®) , leflunomide(Arthfree®) , hydroxychloroquine (plaquenil®) and sulfasalazine(colosalazine®) .

SUMMARY:
This study aims to evaluate the effect of l-carnitine as add- on therapy for improving the outcome in rheumatoid arthritis patients.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is an inflammatory autoimmune disease that affects joints of hand, wrist and foot. Its epidemiology is more pronounced in female to male in ratio 3:1 . Etiology of the disease is related to genetics and environmental factors that lead to formation of epitopes initiating autoimmune response . It is characterized by symmetrical polyarthritis in equal or more than 5 joints and it is known that long term inflammation leads to bone deformities, cartilage damage and synovitis. signs and symptoms include pain and tenderness of joints, morning stiffness for more than 30 minutes, fever, fatigue and weight loss . Also, there are extra-articular manifestations like rheumatoid nodules , interstitial lung disease and ocular manifestations like scleritis . Many treatment approaches in RA are based on anti- inflammatory, anti-oxidant and immune suppressive drugs mainly DMARDs. Up till now, there is no anti-inflammatory agent that is both safe and effective equivalent to DMARDs which are first line of treatment and that can be a scientific gap that should be filled in future research prespectives.

L-Carnitine is a nutritional supplement that is used for enhancing performance in

exercises, valproic acid toxicity, Rett syndrome and in case of secondary carnitine deficiency like in end stage renal disease (ESRD). Physiologically, it is synthesized from lysine and methionine. It is involved in energy production by assisting in transportation of long chain fatty acid into the mitochondria where they undergo beta oxidation for ATP production. Several studies have successfully proven that it has antioxidant effect by activating PPAR gamma which is transcription factor that directly increases expression of antioxidant enzymes like super oxide dismutase (SOD) . LC also have anti-inflammatory effect by acting on PPAR gamma that also inhibits Nf-KB pathway, thus decreasing release of inflammatory mediators. That was mentioned in literature done on inflammatory diseases like coronary artery disease and sepsis . The need for an add on therapy in RA increases to improve response to treatment and provide cost effectiveness benefit that opens the door for repurposing trials.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-60 years old
* diagnosed of rheumatoid arthritis according to 2010 American College of Rheumatology/European League Against Rheumatism criteria for at least 6 months
* enrolled patients treated with one of more of conventional DMARDs for ≥ 6 months with stable dose for ≥ 1 month before start of the study
* active RA despite conventional DMARDs treatment (DAS28 ESR more than or equal 3.2)
* patient or legal representative should sign informed consent

Exclusion Criteria:

* pregnant or lactating female
* patients with liver dysfunction (>1.5x the upper limit of normal value for ALT & AST)
* Patients with kidney dysfunction (serum creatinine more than 1.2 mg/dl)
* Patients with any active infection or concurrent malignancy
* patients with uncontrolled medical conditions or other rheumatic diseases
* patients currently taking drugs that could interact with carnitine like: warfarin

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
change in DAS28 ESR for both arms | From enrollment to the end of trial at 12 weeks
  DAS 28-ESR is a score used to measure disease activity in RA patients. it is calculated using an equation where number of tender joints ( out of 28 joints) , number of swollen joints ( out of 28 joints) , patient assessment of disease activity ( using visual analogue scale from zero to 10) and ESR level are used as inputs to give DAS 28-ESR as output . the score will be measured to all participants both at baseline and at end of study. Higher scores indicate higher disease activity .

SECONDARY OUTCOMES:
proportion of patients achieving ACR50% in both arms | From enrollment to the end of trial at 12 weeks
  It is a score used to measure disease activity in RA patients. ACR 50% is achieved when patient have 50% improvement in tender and swollen joints count and three out of the following five : ESR level , patient assessment of disease activity ( using visual analogue scale from 0 to 10) , physician assessment of disease activity ( using visual analogue scale from 0 to 10) , pain assessment ( using visual analogue scale from 0 to 10) and health assessment questionnaire . this outcome will be assessed at end of trial.
change in HAQ DI for both arms | From enrollment to the end of trial at 12 weeks
  HAQ DI stands for health assessment questionnaire disability index that is used to reflect quality of life and functional disability where scores will vary from 0 to 3 and higher scores indicate more disability .
  A validated Arabic copy will be used and measured both at baseline and at end of trial.
change in TNF aplha for both arms | From enrollment to the end of trial at 12 weeks
  anti inflammatory marker
change in MDA for both arms | From enrollment to the end of trial at 12 weeks
  It is an oxidative stress marker where higher values indicates more oxidative stress
change in TAC for both arms | From enrollment to the end of trial at 12 weeks
  It is an oxidative stress marker where higher values indicate better anti oxidant effect .
safety data for both arms | From enrollment to the end of trial at 12 weeks
  A list of drug related adverse events will be reviewed by patients at each follow up visit ( at end of each month ) and at end of study. It will be expressed as nominal data ( number of patients experienced a certain adverse event versus number of those who don't) .

CONTACTS AND LOCATIONS:
Locations (1):
- Demerdash hospital, Cairo, Demerdash, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fries JF, Spitz P, Kraines RG, Holman HR. Measurement of patient outcome in arthritis. Arthritis Rheum. 1980 Feb;23(2):137-45. doi: 10.1002/art.1780230202. PMID 7362664
- [Background] Smolen JS, Landewe RBM, Bijlsma JWJ, Burmester GR, Dougados M, Kerschbaumer A, McInnes IB, Sepriano A, van Vollenhoven RF, de Wit M, Aletaha D, Aringer M, Askling J, Balsa A, Boers M, den Broeder AA, Buch MH, Buttgereit F, Caporali R, Cardiel MH, De Cock D, Codreanu C, Cutolo M, Edwards CJ, van Eijk-Hustings Y, Emery P, Finckh A, Gossec L, Gottenberg JE, Hetland ML, Huizinga TWJ, Koloumas M, Li Z, Mariette X, Muller-Ladner U, Mysler EF, da Silva JAP, Poor G, Pope JE, Rubbert-Roth A, Ruyssen-Witrand A, Saag KG, Strangfeld A, Takeuchi T, Voshaar M, Westhovens R, van der Heijde D. EULAR recommendations for the management of rheumatoid arthritis with synthetic and biological disease-modifying antirheumatic drugs: 2019 update. Ann Rheum Dis. 2020 Jun;79(6):685-699. doi: 10.1136/annrheumdis-2019-216655. Epub 2020 Jan 22. PMID 31969328
- [Background] Yamanaka H, Tanaka E, Nakajima A, Furuya T, Ikari K, Taniguchi A, Inoue E, Harigai M. A large observational cohort study of rheumatoid arthritis, IORRA: Providing context for today's treatment options. Mod Rheumatol. 2020 Jan;30(1):1-6. doi: 10.1080/14397595.2019.1660028. Epub 2019 Oct 1. PMID 31475852
- [Background] Jiang F, Zhang Z, Zhang Y, Wu J, Yu L, Liu S. L-carnitine ameliorates the liver inflammatory response by regulating carnitine palmitoyltransferase I-dependent PPARgamma signaling. Mol Med Rep. 2016 Feb;13(2):1320-8. doi: 10.3892/mmr.2015.4639. Epub 2015 Dec 4. PMID 26647854
- [Background] Kiziltunc A, Cogalgil S, Cerrahoglu L. Carnitine and antioxidants levels in patients with rheumatoid arthritis. Scand J Rheumatol. 1998;27(6):441-5. doi: 10.1080/030097498442271. PMID 9855215
- [Background] Conforti A, Di Cola I, Pavlych V, Ruscitti P, Berardicurti O, Ursini F, Giacomelli R, Cipriani P. Beyond the joints, the extra-articular manifestations in rheumatoid arthritis. Autoimmun Rev. 2021 Feb;20(2):102735. doi: 10.1016/j.autrev.2020.102735. Epub 2020 Dec 17. PMID 33346115
- [Background] Bongartz T, Nannini C, Medina-Velasquez YF, Achenbach SJ, Crowson CS, Ryu JH, Vassallo R, Gabriel SE, Matteson EL. Incidence and mortality of interstitial lung disease in rheumatoid arthritis: a population-based study. Arthritis Rheum. 2010 Jun;62(6):1583-91. doi: 10.1002/art.27405. PMID 20155830
- [Background] Sayah A, English JC 3rd. Rheumatoid arthritis: a review of the cutaneous manifestations. J Am Acad Dermatol. 2005 Aug;53(2):191-209; quiz 210-2. doi: 10.1016/j.jaad.2004.07.023. PMID 16021111
- [Background] Smolen JS, Aletaha D, McInnes IB. Rheumatoid arthritis. Lancet. 2016 Oct 22;388(10055):2023-2038. doi: 10.1016/S0140-6736(16)30173-8. Epub 2016 May 3. PMID 27156434
- [Background] Klareskog L, Ronnelid J, Saevarsdottir S, Padyukov L, Alfredsson L. The importance of differences; On environment and its interactions with genes and immunity in the causation of rheumatoid arthritis. J Intern Med. 2020 May;287(5):514-533. doi: 10.1111/joim.13058. PMID 32176395
- [Background] Crowson CS, Matteson EL, Myasoedova E, Michet CJ, Ernste FC, Warrington KJ, Davis JM 3rd, Hunder GG, Therneau TM, Gabriel SE. The lifetime risk of adult-onset rheumatoid arthritis and other inflammatory autoimmune rheumatic diseases. Arthritis Rheum. 2011 Mar;63(3):633-9. doi: 10.1002/art.30155. PMID 21360492